CLINICAL TRIAL: NCT02489565
Title: Telemedicine in Qualifying Care Transition Between Tertiary and Primary Health Care Among Stable Coronary Artery Disease Patients: a Randomized Non-inferiority Trial
Brief Title: Telemedicine Qualifying Transition Between Tertiary and Primary Health Care in Stable Coronary Artery Disease Patients
Acronym: Tele_DAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Ministry of Health, Brazil (Other Government); Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: GPPG 14-0206; 401463/2013-3 (Other Grant/Funding Number: MCTI/CNPq/Ministry of Health - SCTIE/DECIT)
Record Dates: First submitted 2015-05-13; First posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; stable; Telemedicine; Patient Discharge
MeSH Terms: conditions — Coronary Artery Disease | interventions — Telemedicine; Primary Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tertiary care (No Intervention): Outpatient from tertiary care with discharge criteria who remains in the tertiary care.
- Primary care (Experimental): Outpatient discharge from tertiary care to a primary care near the patient's home with the support of telemedicine.
  Interventions: Other: Telemedicine

INTERVENTIONS:
Other: Telemedicine — Outpatient discharge from tertiary care to primary care with a letter of referral explaining about the study containing phone number from telemedicine and a letter with the patient's history in the hospital. Two months after discharge, the telemedicine's cardiologist initiates contact with the primary care's physician about patient follow-up.
  Other Names: Primary care with the support of telemedicine
  Arms: Primary care

SUMMARY:
The purpose of this study is to determine whether the telemedicine use in primary health care is effective in the accompaniment of stable coronary artery disease patients who were discharged from the tertiary health care clinics.

DETAILED DESCRIPTION:
This study is a randomized non-inferiority trial for patients with chronic coronary artery disease from a tertiary hospital with outpatient discharge criteria. The purpose is to compare the use of telemedicine in the quality of care transition between tertiary care and primary care patients (intervention group), with patients who remain in the outpatient clinic of a tertiary hospital (control group).

ELIGIBILITY:
Inclusion Criteria:

* individuals with diagnosis of Coronary Artery Disease (CAD) in Canadian Cardiovascular Society (CCS)'s functional classification of angina Class I or II
* patients who did not submit hospitalization for cardiovascular disease in the last year

Exclusion Criteria:

* patients who were not followed up in the health service to at least one year
* unstable patients requiring adjustments of medications or who are performing some diagnostic evaluation at discharge outpatient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants that stay in Canadian Cardiovascular Society (CCS) Functional Classification of Angina I and II as a measure of safety | within one year after discharge
  Not evolve into a higher class than the measure before the intervention

SECONDARY OUTCOMES:
Number of participants with instability of the disease | within one year after discharge
  the need to seek emergency care for cardiovascular disease post intervention.
blood pressure control | within one year after discharge
  verified to maintain systemic blood pressure from the observation of a variation of at least 5% in pre and post intervention measurements
dyslipidemia control | within one year after discharge
  verified to maintain dyslipidemia control through laboratory examination, from the observation of a variation of at least 5% in pre and post intervention measurements of Low Density Lipoproteins (LDL) in blood
diabetes control | within one year after discharge
  verified to maintain diabetes control through laboratory examination, from the observation of a variation of at least 5% in pre and post intervention measurements of fasting glucose in the blood

OTHER OUTCOMES:
Number of participants with control of tobacco | within one year after discharge
  remain without smoking for non smokers; and smoking cessation for smokers
Number of participants in physical activity | within one year after discharge
  maintenance or start regular physical activity post intervention
Access to primary health care | within six months and one year after discharge
  medical consultation in Basic Health Unit held with assessment of current medications and providing prescription.

CONTACTS AND LOCATIONS:
Overall Officials: Carisi A Polanczyk, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Instituto de Avaliação de Tecnologia em Saúde (Institute of Technology Assessment in Health), Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Ruschel KB, Rados DR, Furtado MV, Batista JDL, Katz N, Harzheim E, Polanczyk CA. Transition of care of stable ischaemic heart disease patients from tertiary to primary care with telemedicine support: Randomized noninferiority clinical trial. J Telemed Telecare. 2022 Jan;28(1):52-57. doi: 10.1177/1357633X20906648. Epub 2020 Mar 18. PMID 32188310
- [Derived] Batista Jd, Furtado MV, Katz N, Agostinho MR, Neto BS, Harzheim E, Polanczyk CA. Telemedicine-supported transition of stable coronary artery disease patients from tertiary to primary health care facilities: protocol for a randomized non-inferiority trial. BMC Health Serv Res. 2016 Jul 7;16:227. doi: 10.1186/s12913-016-1469-4. PMID 27387752